CLINICAL TRIAL: NCT01899937
Title: Effect of Different Methodologies on Reliability of Flow Mediated Dilation as Measurement Tool: Meta-regression Analysis to Determine Minimum Quality Standards
Brief Title: Effect of Different Methodologies on Variability of Brachial Artery Flow Mediated Dilation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Top Institute Food and Nutrition (Other)
Responsible Party: Principal Investigator, Lian Engelen, PhD, Maastricht University Medical Center
Other Study IDs: TIFN-CH001-IWG-FMD
Record Dates: First submitted 2013-07-03; First posted 2013-07-16 (Estimated); Last update posted 2013-07-16 (Estimated); Status verified 2013-07

CONDITIONS: Endothelial Dysfunction
Keywords: Endothelial dysfunction; Flow mediated dilation; Brachial artery flow mediated dilation; FMD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

SUMMARY:
Flow mediated dilation (FMD) of the brachial artery has been widely used as a non-invasive measure of endothelial function. FMD independently predicts future cardiovascular events and can be readily influenced by pharmacological, dietary or lifestyle interventions. However, the interpretation of FMD data is currently importantly hampered by differences in measurement methodologies and analysis techniques between laboratories. These differences result in large variation of 'normal' values between laboratories, highlighting the need for adopting widely supported and evidence-based guidelines.

DETAILED DESCRIPTION:
Background: Flow mediated dilation (FMD) of the brachial artery has been widely used as a non-invasive measure of endothelial function. FMD independently predicts future cardiovascular events and can be readily influenced by pharmacological, dietary or lifestyle interventions.

Need for a review: Differences in methodology, guidelines (to control for moderating factors) and analysis techniques contribute to large variation in FMD between laboratories, limiting the widespread use and interpretation of FMD data.

Objectives: To identify methodological and technological factors that contributes to the variability (i.e. repeatability) of the brachial artery FMD. This will allow for development of quality guidelines for FMD measurement based on systematic data analysis.

Design: The planning and conduct of the proposed meta-analyses will follow the Cochrane handbook for systematic reviews of interventions. The reporting will follow the Preferred Reporting Items for Systematic reviews and Meta-Analyses (PRISMA) guidelines.

Data sources: MEDLINE, EMBASE Chemical Abstracts, Biosis and The Cochrane Central Register of Controlled Trials will be searched using appropriate search terms.

Study selection: Observational cohorts and control groups of intervention studies with ≥ 50 subjects.

Methods: A list of quality criteria for scoring of FMD data will be defined both by expert consensus and by thorough review of the literature. Subsequently, a database of brachial artery FMD data (from published data and available individual data) will be compiled. The investigators will investigate which of the quality criteria significantly contribute to the variability of FMD by multiple meta-regression analyses. This data set will also allow us to investigate which quality criteria have the strongest impact on the variability of the FMD, to further refine the list of quality criteria.

ELIGIBILITY:
Inclusion Criteria:

* Observational cohorts and control groups of intervention studies with ≥ 50 subjects

Exclusion Criteria:

* ≤ 50 subjects
* Any co-intervention in control groups of intervention studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults - varied
Sampling Method: Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2013-06; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Brachial artery flow mediated dilation (FMD) analysis | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Ghiadoni, Principal Investigator — University of Pisa; Dick Thijssen, Principal Investigator — Radboud University Medical Center
Locations (4):
- University of Pisa, Pisa, Italy
- Netherlands (3):
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Unilever R&D Vlaardingen, Vlaardingen
  - Top Institute Food and Nutrition, Wageningen